CLINICAL TRIAL: NCT00683046
Title: T-Cell Depleted Allogeneic Stem Cell Transplantation for Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11300A
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myelogenous Leukemia; Lymphoid Leukemia; Chronic Myelogenous Leukemia; Malignant Lymphoma; Hodgkin's Disease; Chronic Lymphocytic Leukemia; Myeloproliferative Disorder; Anemia, Aplastic; Myelodysplastic Syndromes
Keywords: Relapsed or refractory acute myelogenous or lymphoid leukemia.; Acute myeloid or lymphocytic leukemia in first remission at high-risk for recurrence.Chronic myelogenous leukemia in accelerated phase or blast-crisis.; Chronic myelogenous leukemia in chronic phase; Chronic myelogenous leukemia in accelerated phase or blast-crisis; Recurrent or refractory malignant lymphoma or Hodgkin's disease.; Chronic lymphocytic leukemia, relapsed or with poor prognostic features.; Myeloproliferative disorder (polycythemia vera, myelofibrosis) with poor prognostic features.; Severe aplastic anemia after failure of immunosuppressive therapy.; Myelodysplastic syndromes (including PNH); Multiple myeloma at high risk for disease recurrence.
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphoid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Myeloproliferative Disorders; Anemia, Aplastic; Myelodysplastic Syndromes; Recurrence; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis | interventions — fludarabine; Melphalan; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug Intervention (Experimental)
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Stem cells; Drug: Campath

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2 intravenously daily at the same time over 30 minutes on days -7,-6,-5,4,-3,.
Drug: Melphalan — Melphalan 140 mg/m2 IV on day -2.
Drug: Stem cells — Stem cell infusion on day 0.
Drug: Campath — Campath, 20 mg IV on day -7, 6, -5, -4, and -3.

SUMMARY:
Objectives:

1. To evaluate disease free survival after Campath 1H-based in vivo T-cell depletion and non-myelo-ablative ablative stem cell transplantation in patients with hematologic malignancies.
2. To evaluate the incidence and severity of acute and chronic GVHD after Campath 1H-based in vivo T-cell depletion, in patients with hematologic malignancies undergoing non-myelo-ablative stem cell transplantation.
3. To evaluate engraftment and chimerism after Campath 1H-based in vivo T-cell depletion and non-myelo-ablative ablative stem cell transplantation in patients with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Zubrod performance status 2 (See Appendix B).
* Life expectancy is not severely limited by concomitant illness.
* Adequate cardiac and pulmonary function. Patients with decreased LVEF or PFTS will be evaluated by cardiology or pulmonary prior to enrollment on this protocol.
* Serum creatinine <1.5 mg/dL or Creatinine Clearance >50 ml/min .
* Serum bilirubin 2.0 mg/dl, SGPT <3 x upper limit of normal
* No evidence of chronic active hepatitis or cirrhosis.
* HIV-negative
* Patient is not pregnant
* Patient or guardian able to sign informed consent.

Exclusion Criteria:

* N/A

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2001-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Artz, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- T-cell Depleted Allogeneic Stem Cell Transplantation: All patients were administered the following drugs;
  1. Fludarabine 30mg/m2 intravenously daily at the same time over 30 min on days -7,-6,-5,-4, and -3
  2. Melphalan 140mg/m2 IV on day -2
  3. Stem cell infusion on day 0
  4. Campath 20mg IV on day -7,-6,-5,-4, and -3
Period: Overall Study
Arm/Group | T-cell Depleted Allogeneic Stem Cell Transplantation
Started | 204
Completed | 204
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | T-cell Depleted Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 111

OUTCOME MEASURES:

1. Primary Outcome: Median Disease-free Survival
Description: All patients were administered the following drugs;
  1. Fludarabine 30mg/m2 intravenously daily at the same time over 30 min on days -7,-6,-5,-4, and -3
  2. Melphalan 140mg/m2 IV on day -2
  3. Stem cell infusion on day 0
  4. Campath 20mg IV on day -7,-6,-5,-4, and -3
Time Frame: Patients evaluated continuously with disease specific re-evaluation at day 30, 3 months, 6 months, 1 year, and as indicated thereafter up to 10 years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | T-cell Depleted Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 204
Days | 333 [253 to 386]

2. Secondary Outcome: Median Overall Survival
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | T-cell Depleted Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 204
Days | 547 [378 to 946]

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | T-cell Depleted Allogeneic Stem Cell Transplantation
Serious Adverse Events (participants affected / at risk) | 69/204
Other Adverse Events (participants affected / at risk) | 0/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T-cell Depleted Allogeneic Stem Cell Transplantation (N=204)
Abdomial infection (Infections and infestations) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Adult Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 8
Atrial fibrillation (Cardiac disorders) | 2
Bladder infection (Infections and infestations) | 1
Blood and lymphatic system disorders, other (Blood and lymphatic system disorders) | 2
Bone infection (Infections and infestations) | 1
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Catheter related infection (Infections and infestations) | 5
Chronic kidney disease (Renal and urinary disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Confusion (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Endocarditis infective (Cardiac disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Fever (General disorders) | 1
Heart Failure (Cardiac disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Infection and infestations - other, specify (Infections and infestations) | 23
Pharyngitis (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Post operative hemorrhage (Injury, poisoning and procedural complications) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Retinal detachment (Eye disorders) | 1
Sepsis (Infections and infestations) | 11
Skin infection (Infections and infestations) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Syncope (General disorders) | 1
Thromboembolic event (Vascular disorders) | 3
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 4
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No